CLINICAL TRIAL: NCT02924675
Title: Interest of Pregabalin (Lyrica) on the Treatment of Reflex Earache in Head and Neck Cancer.
Acronym: LYRORL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: not sufficiency recruitment
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013_21; 2014-000505-12 (EudraCT Number)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2017-11

CONDITIONS: Earache
Keywords: neuropathic pain, ent cancer, pregabalin
MeSH Terms: conditions — Earache; Neuralgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pregabalin group (Experimental)
  Interventions: Drug: Pregabalin
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — 150mg daily in three doses during three weeks
  Arms: pregabalin group
Drug: Placebo — Three doses daily with lactose
  Arms: Placebo group

SUMMARY:
Referred otalgia is one of the symptoms of oropharynx and hypopharynx cancer. It can be primary (otodynia) or secondary (referred otalgia and projected pain). The mechanism of referred otalgia involves several non adjacent nerve territories as those of head, neck or ear. Referred otalgia is a projected pain due to injury (most of the time cancer) localized far from the ear but sharing the same innervation. In this contest, the otoscopy is normal.

Four cranial nerves participate in the sensory innervation of the external ear: the trigeminal nerve (V) via the auriculo temporal nerve (V3), the facial nerve (VII) for the Ramsay-Hunt's zone with the conch, tragus, antitragus, a part of the anthelix, of the external auditory meatus and of the eardrum, the glossopharyngeal nerve (IX) via the Jacobson's nerve for the external ear canal and the C2 and C3 cervical plexus. However, there are important interindividual anatomical variations.

The relationship between referred otalgia and probable nerve damage has been described. In he oropharynx and hypopharynx, the proximity of the sensory innervation of the ear can then explain the otalgia during the cancer progression. Then referred otalgia has a neuropathic component.

In the literature, the curative treatment of referred otalgia is the cancer treatment. However, the high intensity of referred otalgia leads the patients to a large consumption of analgesics in particular of opioids. These latter are particularly adapted for pain resulting from excess of nociceptive stimulation. Pregabalin (Lyrica®) is an analogue of gamma aminobutyric acid. This molecule binds to alpha subunit 2 delta 1 calcium dependent voltage channels in the central nervous system. its effectiveness has been demonstrated for the treatment of neuropathic pain on diabetic neuropathy, post herpetic neuralgia, lesions in the bone marrow but also the postoperative pain when the molecule is administered after the surgery. The anti hyperalgesic activity of pregabalin is at a dosage of 150mg/day in two or three daily doses.

The purpose of this study was to evaluate the activity of pregabalin administered orally for three weeks after the anesthesia consultation on the intensity of the pain of referred otalgia and on its neuropathic component.

ELIGIBILITY:
Inclusion Criteria:

* referred otalgia
* ENT cancer
* ASA score 1,2 or 3
* understanding protocol
* information and free and informed consent

Exclusion Criteria:

* ASA score 4 et 5
* allergy or intolerance of pregabalin
* creatinin clearance inferior of 50ml/min (Cockcroft formula)
* liver failure
* cardiac failure
* history epilepsy
* ant hyperalgesic treatment
* minor or disabled adult
* intellectual disabilities that prevent the understanding of the protocol
* uncooperative patient
* pregnant women
* patient participating in another research protocol
* lactose intolerant patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-06-05 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
decreased intensity of pain in referred otalgia | three weeks
  diminution of the pain intensity numerical rating scale (NRS)

SECONDARY OUTCOMES:
neuropathic pain | Three weeks
  diminution of the Neuropathic Pain Scale Inventory (NPSI)
Numeric rating Scale | one, three and six months
  referred otalgia after surgery: intensity
Neuropathic Pain Symptom Inventory | one, three and six months
  referred otalgia after surgery: presence

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No